CLINICAL TRIAL: NCT04449601
Title: Comparison of Maternal Neonatal Outcomes of Normotensive and Hypertensive Placental Abruptions: A Novel Approach
Brief Title: Normotensive and Hypertensive Placental Abruptions
Status: Completed | Type: Observational
Sponsor: Hatice Akkaya (Other Government)
Responsible Party: Sponsor-Investigator, Hatice Akkaya, Associate Professor, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Other Study IDs: E52332816/49
Record Dates: First submitted 2020-06-20; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Abruptio Placentae; Affecting Fetus or Newborn
Keywords: Abruptio placenta; complete blood count; hypertension; perinatal outcome.; mean platelet volume
MeSH Terms: conditions — Abruptio Placentae; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (with hypertension ): Two groups were classified regarding of presence or absence of hypertension (53 hypertensive, 62 normotensive).
  Interventions: Other: clinical assesment
- Group 2( without hypertension): Two groups were classified regarding of presence or absence of hypertension (53 hypertensive, 62 normotensive).
  Interventions: Other: clinical assesment

INTERVENTIONS:
Other: clinical assesment — Comparison of Hypertensive group and normotensive group

SUMMARY:
Placental abruption is a significant cause of both maternal morbidity and neonatal morbidity and mortality. Most abruptions accept to be related to a chronic placental disease process. Therefore, it is very important to understand these processes. To analyze maternal and neonatal effects of placental abruption(PA) through a novel classification in the presence of hypertension. Initial hemoglobin parameters were also compared to predict pregnancy outcomes in addition to hypertension.

DETAILED DESCRIPTION:
Objective: We aimed to classify placental abruption according to hypertension status.

Methods: This retrospective cohort designed study was conducted on 115 pregnant women with placental abruption. The main parameters scanned and recorded from the hospital database and patient medical files. Two groups were classified regarding of presence or absence of hypertension (53 hypertensive, 62 normotensive). Maternal demographical and clinical characteristics (abdominal pain, vaginal bleeding) were recorded. APGAR scores below 5 at 1 and 5 min., fetal or neonatal death, admission and length of stay in Neonatal Intensive Care Unit(NICU) were also investigated and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous,
* singleton pregnancies
* above 25 weeks of gestations with positive fetal cardiac activity

Exclusion Criteria:

* multiple gestations,
* presence of fetal or maternal infection,
* chronic inflammatory diseases or connective tissue disorders
* history of myocardial infarction,
* thrombosis
* history of steroid drug usage.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups were formed according to presence or absence of hypertension (53 hypertensive, 62 normotensive) who has placental abruption.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
blood pressure measurement | 2 minute
  mm Hg

SECONDARY OUTCOMES:
hemogram parameters WBC(white blood cell) ,PLT(Platelet), MPV(mean platelet volume), HGB(hemoglobin), Neutrophil lymphocyte ratio..) | first 1 hour
  complete blood test retrospective complete blood count analysis
maternal and newborn length, weight | 5 minute
  centimeters,kilogram
APGAR score | 5 minute
  1st and 5th minute newborn assesment

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Akkaya, Ass Prof, Principal Investigator — Kayseri Education and Research Hospital

IPD SHARING:
Plan to Share IPD: No
The data belonging to participant only will be available to any researcher or editorial review board if needed.